CLINICAL TRIAL: NCT06387212
Title: 35 kDa Hyaluronan Fragment (HA35) Reduces Chronic Skin Inflammation
Brief Title: 35 kDa Hyaluronan Fragment (HA35) Reduces Chronic Inflammation of Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhia Impex LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUI0001
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Skin Inflammation; Cosmetic Skin
Keywords: whitening; pore size; skin dryness; erythema; skin hardness
MeSH Terms: conditions — Dermatitis; Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DermaShine PRO negative microneedles instrument (Experimental)
  Interventions: Drug: 35 kDa hyaluronan fragment HA35 injection

INTERVENTIONS:
Drug: 35 kDa hyaluronan fragment HA35 injection — First, apply an appropriate amount of compound lidocaine cream to the treatment site ( national drug approval number H20063466 ; Beijing Ziguang Pharmaceutical Co., Ltd. ) waited for 60 minutes after applying hemp, and then injected the syringe containing sterile HA35 prepared in advance into the subcutaneous 1.0-1.5mm through the DermaShine PRO negative pressure microneedle importer ( Demasha, South Korea ).
  Other Names: HA35

SUMMARY:
To explore the clinical effect and safety of 35 kDa hyaluronic acid fragment ( HA35 ) combined with negative pressure microneedle technology in improving skin problems.

ELIGIBILITY:
Inclusion Criteria:

* Skin problems include but are not limited to dry skin, dark skin, and coarse pores.
* Chronic skin inflammation, pigmentation, erythema, etc.
* Cooperate with the experimental requirements and be able to complete the score independently。

Exclusion Criteria:

* Pregnant or lactating women.
* Suffering from psychological or mental illness.
* Life is not regular, overeating.
* Hypersensitive to hyaluronic acid, and has a scar constitution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
A skin dryness scale | 120 minutes and 960 minutes
  The Numerical Rating Scale (NRS) was revised and improved, and the 10-point digital score was used to allow the subjects to self-evaluate the skin effect before and after treatment for 120 minutes and 960 minutes. 0 represents no skin dryness, while 10 represents the worst degree of skin dryness.
A fair or smooth skin scale | 120 minutes and 960 minutes
  The Numerical Rating Scale (NRS) was revised and improved, and the 10-point digital score was used to allow the subjects to self-evaluate the skin effect before and after treatment for 120 minutes and 960 minutes. 0 represents the worse degree of fair or smooth skin, while 10 represents the best degree of fair or smooth skin.
A skin pore size scale | 120 minutes and 960 minutes
  The Numerical Rating Scale (NRS) was revised and improved, and the 10-point digital score was used to allow the subjects to self-evaluate the skin effect before and after treatment for 120 minutes and 960 minutes. 0 represents the best degree of skin pore size, while 10 represents the worst degree of skin pore size.
A inflammatory skin thick hardness scale | 120 minutes and 960 minutes
  The Numerical Rating Scale (NRS) was revised and improved, and the 10-point digital score was used to allow the subjects to self-evaluate the skin effect before and after treatment for 120 minutes and 960 minutes. 0 represents the best degree of inflammatory skin thick hardness, while 10 represents the worst degree of inflammatory skin thick hardness.
An erythema color and area scale | 120 minutes and 960 minutes
  The Numerical Rating Scale (NRS) was revised and improved, and the 10-point digital score was used to allow the subjects to self-evaluate the skin effect before and after treatment for 120 minutes and 960 minutes. 0 represents the best degree of erythema color and area, while 10 represents the worst degree of erythema color and area scale.

SECONDARY OUTCOMES:
Self-satisfaction evaluation | 1 week after the end of the treatment
  One week after the end of the treatment, a return visit was conducted to collect the overall satisfaction score of the subjects on the skin treatment. Using the questionnaire (0-10 score) to assess this outcome measure. 0 represents the most dissatisfied, while 10 represents the most satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Nahia Impex LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No